CLINICAL TRIAL: NCT04079725
Title: Histopathological Examination of Iris Tissue in Primary Congenital Glaucoma
Brief Title: Iris Tissue in Primary Congenital Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Abdelkarem Hasan, Resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: primary congenital glaucoma
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Primary Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos | interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental : Infants with primary congenital glaucoma (Experimental)
  Interventions: Procedure: Combined trabeculotomy-trabeculectomy with mitomycin c

INTERVENTIONS:
Procedure: Combined trabeculotomy-trabeculectomy with mitomycin c — Combined trabeculotomy-trabeculectomy with mitomycin C Will be done in all cases then histopathological examination of iris tissue to detect the nature of the disease
  Other Names: Histopathological examination of iris tissue

SUMMARY:
To present the histopathological features of the iris tissue in primary congenital glaucoma which may play a role in pathogenesis

DETAILED DESCRIPTION:
Primary congenital glaucoma etiology still remains obscure . originally barkan , and later Worst , proposed that a membrane covered the anterior chamber angle and blocked aqueous outflow , but the presence of that membrane has not been established histopathologically to date . Now most authors believe that the site of obstruction is the trabecular meshwork rather than an overlying membrane . Maldevelopment of the anterior segment is present in all forms of congenital glaucoma . this maldevelopment may involve the trabecular meshwork alone or the trabecular meshwork in combination with the iris or cornea or both. In approcimately 50% of patients , isolated trabeculodysgensis is the only developmental ocular anomaly found .This is the classic defect found in primary congenital glaucoma .These eyes have no developmental anomalies of iris or cornea present except abnormal insertion of the iris into the angle

ELIGIBILITY:
Inclusion Criteria:

1. Typical symptoms of epiphora , photophobia and blepharospasm
2. corneal diameter > 13 mm
3. Increased ocular tension > 25 mmHg UGA using schiotz tonometer

Exclusion Criteria:

1. Infants with history of previous surgery
2. Secondary glaucoma
3. Glaucoma associated with other congenital anomalies

Ages: 7 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Present histopathological features of iris tissue in infants with primary congenital glaucoma which may play a role in pathogenesis | 2 years
  Histopathological features of iris tissue in infants with primary congenital glaucoma who underwent Combined trabeculotomy-trabeculectomy with mitomycin C

REFERENCES:
- [Background] Mandal AK, Naduvilath TJ, Jayagandan A. Surgical results of combined trabeculotomy-trabeculectomy for developmental glaucoma. Ophthalmology. 1998 Jun;105(6):974-82. doi: 10.1016/S0161-6420(98)96022-5. PMID 9627644
- [Background] Suri F, Yazdani S, Narooie-Nejhad M, Zargar SJ, Paylakhi SH, Zeinali S, Pakravan M, Elahi E. Variable expressivity and high penetrance of CYP1B1 mutations associated with primary congenital glaucoma. Ophthalmology. 2009 Nov;116(11):2101-9. doi: 10.1016/j.ophtha.2009.04.045. Epub 2009 Sep 10. PMID 19744731
- [Background] Biglan AW. Glaucoma in children: are we making progress? J AAPOS. 2006 Feb;10(1):7-21. doi: 10.1016/j.jaapos.2005.10.001. PMID 16527674
- [Background] Black AC, Jones S, Yanovitch TL, Enyedi LB, Stinnett SS, Freedman SF. Latanoprost in pediatric glaucoma--pediatric exposure over a decade. J AAPOS. 2009 Dec;13(6):558-62. doi: 10.1016/j.jaapos.2009.10.003. PMID 20006816
- [Background] Kargi SH, Koc F, Biglan AW, Davis JS. Visual acuity in children with glaucoma. Ophthalmology. 2006 Feb;113(2):229-38. doi: 10.1016/j.ophtha.2005.10.029. Epub 2006 Jan 10. PMID 16406536
- [Background] Mandal AK, Gothwal VK, Bagga H, Nutheti R, Mansoori T. Outcome of surgery on infants younger than 1 month with congenital glaucoma. Ophthalmology. 2003 Oct;110(10):1909-15. doi: 10.1016/S0161-6420(03)00671-7. PMID 14522762
- [Background] Ocular Pathology Atlas. American Academy of Ophthalmology Web site. https://www.aao.org/resident-course/pathology-atlas. Published 2016. Accessed January 4, 2017
- [Background] American Academy of Ophthalmology. Congenital glaucoma, cloudy corneas. https://www.aao.org/image/congenital-glaucoma-cloudy-corneas-2 Accessed July 01, 2019